CLINICAL TRIAL: NCT01669720
Title: BrUOG C261:Single Agent Adjuvant Aflibercept for Patients With Resected or Ablated Metastatic Colorectal Cancer: A Randomized Phase II Study
Brief Title: Adjuvant Aflibercept for Metastatic Colorectal Cancer
Acronym: C261
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy and enrollment
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Lifespan (Other); University of California, San Diego (Other); Montefiore Medical Center (Other); University of Florida (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG C261
Record Dates: First submitted 2012-08-07; First posted 2012-08-21 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic; Colorectal; Colorectal Cancer; Resected or Ablated Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aflibercept (Experimental): Patients will be randomized 2:1, to receive Aflibercept,4mg/kg IV q2weeks until progression for a maximum of 2 years
  Interventions: Drug: Aflibercept
- Observation (No Intervention): Patients will be randomized 2:1 to receive Aflibercept. Patients who are randomized to observation will be followed per the study table, but will receive no intervention.

INTERVENTIONS:
Drug: Aflibercept — Aflibercept: 4mg/kg IV q2weeks until progression for a maximum of 2 years
  Arms: Aflibercept

SUMMARY:
The main purpose of this study is to evaluate if aflibercept can reduce the chance that metastatic (spread of) colorectal cancer can grow back after finishing standard treatment. The study will also look at the side effects of aflibercept and the effect on quality of life.

DETAILED DESCRIPTION:
There are over 1.2 million new cases of colorectal cancer and 600,000 deaths worldwide. The liver is the dominant site of metastases. Approximately 20-25% of patients with advanced colorectal cancer will be candidates for resection/ablation of all sites of metastatic disease.1 Unfortunately, despite resection/ablation of all metastatic sites only about 20% of these patients are ultimately cured.1 An effective adjuvant agent would prevent tumor recurrence.

Aflibercept and bevacizumab are effective when combined with FOLFIRI for metastatic colon cancer. Neither has been tested in a randomized study in the adjuvant setting for patients with resected metastatic disease. Since aflibercept more effectively inhibits all forms of VEGF including VEGF-A, VEGF-B and PIGF, in striking contrast to bevacizumab which inhibits only VEGF-A, aflibercept likely will be more effective than bevacizumab as a single agent in the adjuvant metastatic setting. Therefore, we propose a randomized study of adjuvant aflibercept for patients metastatic colorectal cancer who have received 10-12 cycles of perioperative FOLFOX and have had had a complete response to all sites of metastases after chemotherapy and local modalities such as surgical resection or ablation. SBRT may also be used to produce a complete response in a metastatic site not easily amenable to surgery or ablation. Only patients with very high risk of recurrence, defined as 3 or more metastatic sites, will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 First-line treatment of metastatic colorectal cancer with 3 or more metastases 3.1.2At least 10 cycles of combination therapy with an oxaliplatin or irinotecan based regimen per institutional preference (patients may receive 6 cycles, go to surgery, then complete 4 cycles, they may complete all 10 (or more) prior to surgery, or receive any combination as long as they receive at least 10 cycles. ) 3.1.3 Resection or ablation of all metastatic sites that have not achieved complete response with perioperative therapy (regimen). The sequencing of resection, ablation, and 10-12 cycles of combination therapy (regimen) with an oxaliplatin or irinotecan based regimen may be performed according to standard institutional procedure.

3.1.4 Patients achieving a complete response in a metastatic site by stereotactic body radiation are eligible if the site was not easily accessible by surgery or ablation and a complete response was achieved.

3.1.5 No severe, uncontrolled concurrent illness that would interfere with protocol therapy.

3.1.6 No known CNS disease 3.1.7 ECOG Performance Status 0-2 3.1.8 No chemotherapy or radiation therapy within last 3 weeks 3.1.9 For patients who had 3 months of perioperative therapy (regimen), then surgery, then 3 months of therapy (regimen), patients must be off therapy for no more than 8 weeks prior to randomization. For patients who had all their therapy and then surgery, they must be no more than 8 weeks from surgery prior to randomization.

3.1.10 No concurrent anticancer therapy. 3.1.11 Absolute neutrophil count ≥ 1,500/uL, Hgb > 9.0 g/dl, platelet ≥ 100,000/uL.

3.1.12 Total bilirubin ≤ 1.5x upper limit of normal (ULN) and AST or ALT ≤ 5x ULN; 3.1.13 Creatinine < 1.5 x ULN 3.1.14 Life expectancy of at least 12 weeks. 3.1.15 Age ≥ 18 years 3.1.16 Women of childbearing potential must have a negative pregnancy test. 3.1.17 Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

3.1.18 Voluntary written informed consent.

Exclusion Criteria:

3.2.1 Residual metastatic disease after resection/ablation 3.2.2 Clinically significant cardiac disease (e.g., uncontrolled hypertension [blood pressure of >160/90 mmHg on medication], history of myocardial infarction within 6 months,), New York Heart Association (NYHA) Class II or greater congestive heart failure within 6 months, unstable arrhythmia. Patients with an atrial arrhythmia must have this condition well controlled on stable medication. Patients with current or recent (within 6 months) unstable angina are also not eligible. Documentation of cardiac medical history to be provided.

3.2.3 Significant bleeding diathesis or coagulopathy 3.2.4 History of cerebral aneurysms or cerebral arteriovenous malformations. 3.2.5 Patients with recent (within 12 months) arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), or clinically significant peripheral artery disease should also be excluded.

3.2.6 Patients with a history of a gastrointestinal fistula or perforation. 3.2.7 Women who are breast-feeding. 3.2.8 Patients who have undergone major surgery, chemotherapy, or radiotherapy within the last 3 weeks.

3.2.9 Patients on concurrent anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital (East Greenwich and Newport), Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aflibercept | Observation
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept | Observation | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 9
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [46 to 61] | 57 [44 to 75] | 54.6 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Progressed
Description: Disease free survival in patients with advanced colorectal cancer who have undergone resection/ablation of all metastatic sites.
Time Frame: Every 3 months until disease progression (for up to 2 years).
Measure: Number; unit: participants
Arm/Group | Aflibercept | Observation
Number analyzed (Participants) | 7 | 3
participants | 2 | 0

2. Secondary Outcome: Number of Participants Who Experienced a Toxicity Profile of Adjuvant Ziv-aflibercept, up to 2-years of Duration, for Patients Who Previously Received Systemic Perioperative Therapy (Regimen) and Surgical Resection/Ablation.
Description: Toxicity defined by CTCAE Version 4.0 toxicities
Time Frame: Throughout study treatment until 30 days post off study, approximately 2 years
Population: Data table reflects total number of patients who experienced a toxicity on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept | Observation
Number analyzed (Participants) | 7 | 3
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: Every 2 weeks until 30 days post last dose of drug
Arm/Group | Aflibercept | Observation
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 6/7 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=7) | Observation (N=3)
HTN (Investigations) | 6 (6) | 1 (1)
Bronchial infection (Investigations) | 1 (1) | 0 (0)
UTI (Investigations) | 1 (1) | 0 (0)
ALK (Investigations) | 4 (4) | 0 (0)
Glu (Investigations) | 6 (6) | 0 (0)
proteinuria (Investigations) | 2 (2) | 0 (0)
PLT (Investigations) | 1 (1) | 1 (1)
AST (Investigations) | 3 (3) | 1 (1)
ALT (Investigations) | 2 (2) | 1 (1)
bruising (Investigations) | 1 (1) | 0 (0)
Hoarseness (Investigations) | 2 (2) | 0 (0)
akathisia/restlessness (Investigations) | 1 (1) | 0 (0)
cough (Investigations) | 1 (1) | 0 (0)
fever (Investigations) | 1 (1) | 0 (0)
rash (Investigations) | 1 (1) | 0 (0)
Anemia (Investigations) | 2 (2) | 0 (0)
fatigue (Investigations) | 2 (2) | 0 (0)
lymph (Investigations) | 3 (3) | 0 (0)
Sodium (Investigations) | 3 (3) | 0 (0)
Edema- localized (Investigations) | 2 (2) | 0 (0)
pain-hip/leg, mouth, abd (Investigations) | 5 (5) | 0 (0)
headache (Investigations) | 2 (2) | 0 (0)
mucositis (Investigations) | 1 (1) | 0 (0)
creatinine (Investigations) | 1 (1) | 0 (0)
WBC (Investigations) | 2 (2) | 0 (0)
dizziness (Investigations) | 1 (1) | 0 (0)
neuropathy (Investigations) | 2 (2) | 0 (0)
arthralgia (Investigations) | 1 (1) | 0 (0)
weight gain (Investigations) | 1 (1) | 0 (0)
constipation (Investigations) | 1 (1) | 0 (0)
vision-blurry (Investigations) | 1 (1) | 0 (0)
increased hemoglobin (Investigations) | 1 (1) | 0 (0)
insomnia (Investigations) | 1 (1) | 0 (0)
anorexia (Investigations) | 1 (1) | 0 (0)
Anxiety (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No